CLINICAL TRIAL: NCT04684784
Title: Effect of Dry Needling on Surface Electromyographic Activity in Latent Trigger Points
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Castilla-La Mancha (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DNEMG
Record Dates: First submitted 2020-12-21; First posted 2020-12-28 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2020-12

CONDITIONS: Trigger Point Pain, Myofascial
Keywords: Dry needling; Electromyography; Latent trigger point
MeSH Terms: conditions — Myofascial Pain Syndromes

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Deep Dry Needling (Experimental): Intervention-Dry Needling: Deep Dry Needing into the latent trigger point of the upper trapezius muscle
  Interventions: Device: Intervention-Dry Needling
- Sham Dry Needling (Placebo Comparator): Control-Dry Needling: Sham Dry Needling into the latent trigger point of the upper trapezius muscle
  Interventions: Device: Control-Dry Needling

INTERVENTIONS:
Device: Intervention-Dry Needling — Deep Dry Needling into the site of the latent TriggerPoint of the upper trapezius muscle. 1 session in upper trapezius muscle moving the needle up and down ten times.
  Arms: Deep Dry Needling
Device: Control-Dry Needling — Sham Dry Needling into the site of the latent Trigger Point of the upper trapezius muscle with non-penetrating needles
  Arms: Sham Dry Needling

SUMMARY:
Brief summary: The purpose of this study is to determine the effect of Dry Needling (DN) on electromyographic activity in different situations at the latent trigger point (LTrP) point of the upper trapezius. Randomized controlled trial, in parallel with the crossover control design. Two groups with LTrP in the upper trapezius, and the DN group or the Sham-Dn group will be randomly selected.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 30 years
* The presence of LTrP in the middle third of the upper trapezius muscle onthe dominant side
* Being able to provide written informed consent
* Being able to follow instructions and realize clinical tests

Exclusion Criteria:

* Any pharmacological therapeutic
* Any medical treatment or physical therapies at cervical region during the 6-month before this study
* Any diagnosed health problem
* Any history of head and upper extremity surgery or trauma
* Any red flags to DN, (ie: metabolic diseases, pregnancy, kinesiophobia,Infection, cancer)• Absence of recurrent history of neck pain
* No neck pain symptomatology the previous 6 months
* Cervical disk herniation

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2021-01-04 (Actual); Primary Completion 2021-02-04 (Actual); Study Completion 2021-02-18 (Actual)

PRIMARY OUTCOMES:
Changes in resting surface EMG activity (amplitude, RMS) | Baseline, at 30 minutes after treatment, at 24 hours after treatment, at 72 hours after treatment
  EMG activity (RMS) of the upper trapezius after dry needling or sham needling as assessed by the EMG ME 6000 TE(Mega Electronics, Kuopio, Finland). Resting EMG activity will be expressed as a percentage of maximal reference contractions of the upper trapezius (% reference contractions).

SECONDARY OUTCOMES:
Changes in resting surface EMG activity (Median frequency, MF) | Baseline, at 30 minutes after treatment, at 24 hours after treatment, at 72 hours after treatment
  EMG activity (RMS) of the upper trapezius after dry needling or sham needling as assessed by the EMG ME 6000 TE(Mega Electronics, Kuopio, Finland).
  EMG median frequency will be used to determine the endurance of the upper trapezius. The EMG median frequency will be measured in Hertz (Hz).
Changes in submaximal contrations surface EMG activity of upper trapezius (amplitude, RMS) | Baseline, at 30 minutes after treatment, at 24 hours after treatment, at 7submaximal contractions EMG activity will be expressed as a percentage of maximal reference contractions of the upper trapezius (% reference contractions).2 hours after treatment
  EMG activity (RMS) of the upper trapezius after dry needling or sham needling as assessed by the EMG ME 6000 TE(Mega Electronics, Kuopio, Finland).
  EMG activity of submaximal contractions will be expressed as a percentage of submaximal reference contractions of the upper trapezius (% reference contractions).
Changes in submaximal contrations surface EMG activity of upper trapezius (Median frequency, MF) | Baseline, at 30 minutes after treatment, at 24 hours after treatment, at 72 hours after treatment
  EMG activity (RMS) of the upper trapezius after dry needling or sham needling as assessed by the EMG ME 6000 TE(Mega Electronics, Kuopio, Finland).
  EMG median frequency will be used to determine the endurance of the upper trapezius. The EMG median frequency will be measured in Hertz (Hz).
Change in Pain Pressure Threshold (PPT) | Baseline, at 30 minutes after treatment, at 24 hours after treatment, at 72 hours after treatment
  Pressure-Pain Threshold as assessed by an manual mechanical algometer. PPT is the minimal amount of pressure that produces pain and is used to assess abnormalities in nociceptive processing or hyperalgesia.

CONTACTS AND LOCATIONS:
Overall Officials: Javier Abián-Vicén, PhD, Study Director — University of Castilla-La Mancha
Locations (1):
- Performance and Sport Rehabilitation Laboratory, Toledo, Spain

IPD SHARING:
Plan to Share IPD: No